CLINICAL TRIAL: NCT02958943
Title: Electronic Alert-Based Computerized Decision Support to Increase Prescription of Anticoagulation in High-Risk Atrial Fibrillation Patients in the Outpatient Setting (AF-ALERT2)
Brief Title: Electronic Alerts for Stroke Prevention in Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Samuel Z.Goldhaber, MD, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016D005336
Record Dates: First submitted 2016-11-05; First posted 2016-11-08 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: atrial fibrillation; stroke; computerized decision support
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic Alert (Experimental): Each provider in the alert group will receive an on-screen notification regarding the patient's increased risk of stroke in AF and the lack of an active order for anticoagulation.
  Interventions: Behavioral: On-screen electronic alert
- No Alert (No Intervention): Each provider in the non-alert group will receive no such notification.

INTERVENTIONS:
Behavioral: On-screen electronic alert — On-screen notification regarding the patient's increased risk of stroke in AF and the lack of an active order for anticoagulation. Providers may then 1) access a template of FDA-approved anticoagulation regimens for stroke prevention in AF, 2) follow a link to evidence based clinical practice guidelines, or 3) proceed onto order entry after providing an explanation for why anticoagulation was not prescribed.
  Arms: Electronic Alert

SUMMARY:
Atrial fibrillation (AF) is the most preventable cause of stroke. However, despite widely available risk stratification tools, five options for oral anticoagulation, and evidence-based practice guidelines, anticoagulation for stroke prevention in AF is consistently under-prescribed. Data from this center (Brigham and Women's Hospital [BWH]) (1) demonstrate that fewer than 50% of outpatients with AF at high-risk for stroke according to 2012 Focused Update of the European Society of Cardiology Guidelines for the Management of AF (2) receive anticoagulation.

Aim #1: To determine the impact of electronic alert-based computerized decision support (CDS) on prescription of anticoagulation in high-risk AF patients in the outpatient setting who are not being prescribed anticoagulation for stroke prevention.

Hypothesis #1: Electronic alert-based CDS will increase prescription of anticoagulation by 80% in high-risk AF patients in the outpatient setting who are not being prescribed anticoagulation for stroke prevention.

Aim #2: To determine the impact of electronic alert-based computerized decision support (CDS) on the frequency of stroke and systemic embolic events in high-risk AF patients in the outpatient setting who are not being prescribed anticoagulation for stroke prevention.

Hypothesis #2: Electronic alert-based CDS will reduce the frequency of stroke and systemic embolism in high-risk AF patients in the outpatient setting who are not being prescribed anticoagulation for stroke prevention. Data acquired through this study regarding the frequency of stroke and systemic embolism will be used to calculate sample size requirements for a future clinical end-point driven randomized controlled trial of electronic alerts to prevent stroke in high-risk AF patients.

DETAILED DESCRIPTION:
AF is associated with an increased risk of fatal and disabling ischemic stroke. Despite widely accessible evidence-based clinical practice guidelines, risk stratification tools (CHA2DS2-VASc and HAS-BLED) and five effective oral antithrombotic agents for stroke prevention (22), at least 40% of high-risk patients with AF worldwide remain unprotected because of failure to prescribe anticoagulation. The failure to prevent stroke in AF has become a critical international patient safety crisis. The root causes of underutilization include lack of provider and patient education about the importance of stroke prevention in AF, inadequate risk stratification, and concerns regarding the bleeding risk with anticoagulant therapy. The investigators were surprised to learn that even at BWH, underutilization of anticoagulation for stroke prevention in AF continues to be a concern (1).

The failure to prevent stroke in AF is similar to the crisis in VTE prevention among hospitalized patients from a decade ago. To address this critical patient safety problem, investigators evaluated the impact of alert-based CDS on VTE prevention (18). First, investigators designed software linked to our Electronic Health Record (EHR) and provider order entry program to identify hospitalized patients at risk for VTE using a weighted risk score and for whom prophylaxis was not ordered. Patients were randomized to the intervention group, in which the responsible physician received an electronic alert regarding the risk of VTE and recommendation regarding prophylaxis, or to the control group, in which no alert was issued. Compared with the control group, electronic alerts more than doubled the rate of thromboprophylaxis orders (from 14.5% to 33.5%; p<0.0001). The risk of symptomatic VTE was reduced by 41% (hazard ratio, 0.59; 95% confidence interval 0.43-0.81; p=0.001) among patients for whom an electronic alert was issued. Investigators have also shown that "human" (person-to-person) alert-based decision support for the prevention of VTE in at-risk hospitalized patients more than doubled the rate of VTE prophylaxis compared with controls during hospitalization (21) and after discharge (19).

The current study will determine the impact of electronic alert-based CDS on prescription of anticoagulation in high-risk AF patients in the outpatient setting who are not being prescribed anticoagulation for stroke prevention. Because this is a Quality Improvement initiative, investigators will not mandate a specific antithrombotic agent, regimen, or duration. Investigators will provide options for anticoagulation to prevent stroke in AF and allow the provider to make the best choice based on their clinical judgment. If there is a contraindication to anticoagulation or if the risks outweigh the benefits of antithrombotic therapy, the provider can elect to omit anticoagulation but will need to provide the rationale for doing so. The current study will also determine the impact of electronic alert-based CDS on the frequency of stroke and systemic embolic events in high-risk AF patients in the outpatient setting who are not being prescribed anticoagulation for stroke prevention. Data acquired through this study regarding the frequency of stroke and systemic embolism will be used to calculate sample size requirements for a future clinical end-point driven randomized controlled trial of electronic alerts to prevent stroke in high-risk AF patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age ≥ 18 years
* Problem list entry of AF or atrial flutter
* CHA2DS2VASc score ≥2

Exclusion Criteria:

* Active prescription for anticoagulant therapy
* CHA2DS2VASc score <2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 798 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
frequency of prescription of anticoagulation in high-risk AF patients in the outpatient setting who are not being prescribed anticoagulation | 48 hours
  frequency of prescription of anticoagulation in high-risk AF patients in the outpatient setting who are not being prescribed anticoagulation for stroke prevention before study randomization. The primary efficacy outcome will be determined by review of the EHR medication documentation for prescription of anticoagulation by 48 hours after randomization.

SECONDARY OUTCOMES:
frequency of stroke/TIA, systemic embolism, myocardial infarction and all-cause mortality | 3 months
  frequency of stroke/TIA, systemic embolism, myocardial infarction and all-cause mortality at 3 months from randomization
frequency of major bleeding (as defined by the ISTH bleeding classification system) | 3 months
  major bleeding (as defined by the ISTH bleeding classification system) at 3 months from randomization

OTHER OUTCOMES:
frequency of stroke, TIA, systemic embolism | 3 months
  frequency of stroke, TIA, systemic embolism
frequency of myocardial infarction | 3 months
  frequency of myocardial infarction
frequency of all-cause mortality | 3 months
  frequency of all-cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Piazza G, Hurwitz S, Campia U, Bikdeli B, Lou J, Khairani CD, Bejjani A, Snyder JE, Pfeferman M, Barns B, Rizzo S, Glezer A, Goldhaber SZ. Electronic alerts for ambulatory patients with atrial fibrillation not prescribed anticoagulation: A randomized, controlled trial (AF-ALERT2). Thromb Res. 2023 Jul;227:1-7. doi: 10.1016/j.thromres.2023.05.006. Epub 2023 May 11. PMID 37182298